CLINICAL TRIAL: NCT02105350
Title: A Phase I Trial of MEK Inhibitor MEK 162 Combined Sequentially With Gemcitabine-Oxaliplatin (GEMOX) in Patients With Advanced Biliary Cancer
Brief Title: A Study of MEK162 With Gemcitabine and Oxaliplatin in Biliary Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was never initiated
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Biliary GEMOX / MEK
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Biliary Tract Carcinoma; Gallbladder Carcinoma
Keywords: MEK162; Gemcitabine; Oxaliplatin; Non-resectable; Recurrent or metastatic
MeSH Terms: conditions — Gallbladder Neoplasms; Recurrence; Neoplasm Metastasis | interventions — Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MEK 162, gemcitabine, and oxaliplatin (Experimental): MEK 162 (30 mg or 45 mg by mouth), twice a day, every day. Gemcitabine (1000 mg/m2 by vein), followed by oxaliplatin (85 mg/m2 by vein) every 2 weeks.
  Interventions: Drug: MEK 162; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: MEK 162
Drug: Gemcitabine
  Other Names: Gemzar
Drug: Oxaliplatin
  Other Names: Eloxatin

SUMMARY:
This is a phase I study (an early study to check the safety of a new drug or drug combination) to find the safest and most tolerated dose of the combination of oxaliplatin with gemcitabine and MEK 162 in patients with biliary cancer (including gallbladder cancers and cancers associated with the bile ducts leading from the gallbladder and to and from the liver) that is not curable by surgery and/or has spread beyond the biliary tree (place where cancer started). Everyone will receive the same standard doses of oxaliplatin and gemcitabine but may receive different doses of MEK 162.

MEK 162 is a new drug which plays an important role in the regulation of cell growth and has been shown to shrink tumours in patients with biliary cancer and other types of human cancers. This type of drug has also been shown to shrink tumours when given in combination with cisplatin and gemcitabine in research studies done in animals and in some patients with biliary cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological or cytological diagnosis of non-resectable, recurrent or metastatic biliary tract (intra- or extra-hepatic) or gallbladder carcinoma.
* Have measurable disease.
* Not received prior systemic therapy for advanced biliary cancer.
* Age 18 years of age or older.
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2.
* Estimated life expectancy is greater than 3 months.
* Have adequate hematological function.
* Have adequate cardiac function.
* All radiology studies performed within 4 weeks prior to the start of therapy.
* No evidence of active uncontrolled infection.
* Ability to understand and willing to sign a written informed consent document.
* Ongoing prior toxicities related to previous treatments received to grade 1 or less at time of registration.
* Able to take oral medications.

Exclusion Criteria:

* Progressing within 6 months of receiving adjuvant treatment for biliary tract cancer.
* Not have received prior chemotherapy for non-resectable or metastatic disease or MEK inhibitor.
* Histopathological or cytological diagnosis of ampullary carcinoma.
* Incomplete recovery from previous surgery.
* Undergoing current treatment with curative intent.
* History of prior malignancy that could interfere with the response evaluation.
* Any evidence of severe or uncontrolled systemic diseases or laboratory findings that may affect participation in the trial.
* Any psychiatric or other disorder likely to impact on informed consent.
* Pregnant or nursing (lactating) women.
* Agree to use highly effective methods of contraception throughout the study and for 6 months after study drug discontinuation.
* Significant cardiac disease.
* History of retinal degenerative disease.
* History of Gilbert's syndrome.
* Known positive serology for HIV, active hepatitis B, and/or active hepatitis C infection.
* Neuromuscular disorders that are associated with elevated creatine kinase.
* Planning on embarking on a new strenuous exercise regimen after first dose of study treatment.
* Impairment of gastrointestinal function or gastrointestinal disease.
* Any other condition that would contraindicate participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Total incidence of grade 3 and 4 adverse events | 2 years
Total rate of grade 3 and 4 adverse events | 2 years
Maximum dose level at which 0/3 patients or 1/6 patients experience dose-limiting toxicity | 2 years

SECONDARY OUTCOMES:
Number of patients with objective response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Knox, M.D., Principal Investigator — Princess Margaret Cancer Centre